CLINICAL TRIAL: NCT05358015
Title: Vascularised Bone Grafts for Treatment of Scaphoid Nonunion: a Case Series Study
Brief Title: Vascularized Bone Grafts for Treatment of Scaphoid Nonunion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa abdelhady Ismail, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBGs for scaphoid nonunion
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Scaphoid Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- scaphoid nonunion (Experimental): pedicled and free ABG for treatment of scaphoid nonunion
  Interventions: Procedure: vascularized bone graft for scaphois nonunion

INTERVENTIONS:
Procedure: vascularized bone graft for scaphois nonunion — vascularized bone graft for scaphois nonunion

SUMMARY:
To assess the effect of vascularized bone grafting on the functional, clinical and radiological outcomes of the scaphoid nonunion

DETAILED DESCRIPTION:
The scaphoid is the most commonly fractured carpal bone accounting for 60% of fractures. A number of case series have identified a 10%-15% nonunion rate. Scaphoid nonunion refers to a spectrum of failed healing, each of which requires a tailored approach.

Subsequent to non-union, degenerative changes with the formation of cysts, bony resorption with loss of bone stock and the development of apex dorsal angulation or the humpback deformity may occur leading to scaphoid non-union advanced collapse (SNAC) of the wrist and the formation of a proximal pole which extends with the lunate.

This has serious functional implications for the patient in terms of wrist range of movement, grip strength and general activities of daily living . The management of nonunion has remained controversial since the last century.

Bone grafting has been performed since the late 1920s with positive results. The importance of vascularity was enforced by finding that in the presence of avascular necrosis ( AVN ), conventional non vascularized bone grafts ( NVBGs) could only achieve a 47% union rate . However, in the absence of AVN, these NVBGs could achieve union rates of 94% .

There was growing consensus that new techniques were required to address the shortfall, and accordingly, vascularized bone grafting (VBG) techniques stemmed from this. It was widely believed that providing adequate blood flow would help treat cases of non-union . Several studies demonstrate that VBGs accelerated bone healing by preserving osteocytes and preventing the slower creeping substitution and were able to increase blood flow and superior mechanical properties in VBGs as opposed to NVBGs . VBGs could be further classified into pedicled or free VBGs. Pedicled VBGs involve isolating a segment of bone local to the defect and maintaining the blood supply to this segment of donor bone which is then fixed into the recipient site. This requires a good stock of donor bone in close proximity to the defect. Free VBGs involve detaching a segment of bone with its vascular bundle from a donor site and anastomosing this to recipient vessels with the fixation of the donor bone to recipient bone.This study hypothesis that VBGs should be used in all cases of humpback deformity , proximal pole fracture , AVN and cystic degeneration from the start.

ELIGIBILITY:
Inclusion Criteria:

All Patients will be included if they met the following criteria:

* Age: all patient more than 18 years up to 55 years
* Fracture: nonunion and a vascular necrosis proved by MRI (Herbert stage I or II) , humpback deformity, Proximal pole fracture, cystic degeneration, failed previous surgery (K wire, Herbert, plate distal radius)
* Pain: persistent disabling pain and tenderness at wrist joint due to scaphoid nonunion.

patient: both sex will included, both handiness, good bone quality.

Exclusion Criteria:

* Commuted Other carpus fractures
* Nonunion less than 3 months
* Radio-carpal Arthritis or instability

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Disability of the arm,shoulder and hand ( DASH) score ranging from 0 to 29 | 2 years
  The final end results will be assessed according to DASH score , a DASH score ranging from 0 to 29 was thought by most respondents to be the point where patients/clients were 'no longer considering their upper-limb disorder a problem .
Mayo wrist score of 60 - 100 will be satisfactory | 2 years
  The final end results will be assessed according to modified Mayo wrist score of 60 - 100 will be satisfactory .
  Secondary (subsidiary):

SECONDARY OUTCOMES:
Carpal Alignment Before and After VBG | 2 years
  the articular surfaces of the proximal and distal carpal rows should form three smooth arcs , the spacing between all carpal bones should be 1-2 mm in antroposterior view and the distal radius, lunate and capitate should be in a straight line in lateral view
Scaphoid Height-to-length ratio | 2 years
  The mean normal H/L ratio in the sagittal plane was 0.61 (range, 0.54-0.69) and in the coronal plane 0.42 (range, 0.36-0.48).
Scapholunate angle | 2 years
  Scapholunate angle is the angle between longitudinal axes of lunate and scaphoid (tangential line from the dorsum of scaphoid) in the lateral radiograph the scapholunate angle should be between 30o and 60o in the neutral position
Radio-lunate angle | 2 years
  Radiolunate angle is the angle between the longitudinal axes of radius and lunate in lateral view
Lateral interscaphoid angle | 2 years
  Normal lateral intrascaphoid angle averages 30 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Kotb, M.D, Study Director — Assiut University

REFERENCES:
- [Background] Dias JJ, Brenkel IJ, Finlay DB. Patterns of union in fractures of the waist of the scaphoid. J Bone Joint Surg Br. 1989 Mar;71(2):307-10. doi: 10.1302/0301-620X.71B2.2925752.
- [Background] Szabo RM, Manske D. Displaced fractures of the scaphoid. Clin Orthop Relat Res. 1988 May;(230):30-8. PMID 3284681
- [Background] El-Karef EA. Corrective osteotomy for symptomatic scaphoid malunion. Injury. 2005 Dec;36(12):1440-8. doi: 10.1016/j.injury.2005.09.003. Epub 2005 Oct 27. PMID 16256995
- [Background] Lynch NM, Linscheid RL. Corrective osteotomy for scaphoid malunion: technique and long-term follow-up evaluation. J Hand Surg Am. 1997 Jan;22(1):35-43. doi: 10.1016/S0363-5023(05)80177-7. PMID 9018610